CLINICAL TRIAL: NCT06886789
Title: An Application of SMART Methodology to Optimize an Intervention to Maintain Improvements in Health Behaviors in Under-resourced Patients After Phase II Cardiac Rehabilitation
Brief Title: SMART to Optimize an Intervention to Maintain Health Improvements After Cardiac Rehabilitation
Acronym: EMPOWER ME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of the Director, National Institutes of Health (OD) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HL171158-01A1 (NIH); 1R01HL171158-01A1 (NIH)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Cardiac Rehabilitation
Keywords: Cardiovascular disease; Cardiac rehabilitation; Medication adherence; Weight loss; Weight management; Weight maintenance; Physical activity; Intervention optimization; Sequential, multiple assignment, randomized trials; Digital health
MeSH Terms: conditions — Cardiovascular Diseases; Medication Adherence; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: Sequential, Multiple Assignment, Randomized Trial (SMART)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- First Intervention: Text Messaging, Second Intervention: Continued Text Messaging (Experimental): Participants are first randomized to the low-intensity text messaging intervention. On 3 days/week they receive a text about 1 of the 3 behaviors (weight maintenance or loss, physical activity, and medication adherence) in randomized order with guidance for maintaining or improving these behaviors to reach program-provided goals. The system compares their last week's adherence to the responder criteria. They receive feedback praising adherence and instructions for a theory-driven behavioral strategy (e.g., stimulus control) to increase adherence. Feedback is tailored to the patient's adherence or existence of self-monitoring data. Participants meeting responder criteria after 2 months will continue to receive the text messaging intervention for the next 3 months.
  Interventions: Behavioral: Text Messaging
- First Intervention: Text Messaging, Second Intervention: Low-Intensity Cardiac Rehabilitation (Experimental): Participants receive the text messaging intervention for 2 months. Following their mid-intervention assessment, they are randomized to receive the low-intensity cardiac rehabilitation maintenance program. Patients are instructed to log in 3 times weekly to view lessons, sync their Fitbit data, and complete a home-based workout video. They track weight, PA, and medication adherence daily. Patients have access to an extensive CR resource library made and curated by the platform provider plus resources on maintaining heart healthy behaviors during Phase III created by the research team. They are reminded to log in if they log in less than twice weekly.
  Interventions: Behavioral: Text Messaging; Behavioral: Low-Intensity Cardiac Rehabilitation Maintenance Program
- First Intervention: Text Messaging, Second Intervention: High-Intensity Cardiac Rehabilitation (Experimental): Participants receive the text messaging intervention for 2 months. Following their mid-intervention assessment, they are randomized to receive the high-intensity cardiac rehabilitation maintenance program. Patients are instructed to log in 3 times weekly to view lessons, sync their Fitbit data, and complete a home-based workout video. They track weight, PA, and medication adherence daily and attend a once weekly virtual meeting with a CR case manager. Meetings are modeled after Phase II and focus on tailored exercise prescription, addressing cognitive, behavioral, and environmental adherence barriers, and support. Patients have access to an extensive CR resource library made and curated by the platform provider plus resources on maintaining heart healthy behaviors during Phase III created by the research team. They are reminded to log in if they log in less than twice weekly.
  Interventions: Behavioral: Text Messaging; Behavioral: High Intensity Cardiac Rehabilitation Maintenance Program
- First Intervention: Fully Automated Online Program (FAOP), Second Intervention: Continued FAOP (Experimental): Patients receiving the fully automated online program will select a weight loss or a weight maintenance curriculum based on their goals. Patients will receive 8 weeks of fully automated lessons covering the 3 key behaviors: weight (management or loss), physical activity, and medication adherence. All 3 behaviors are discussed weekly, but the lessons first prioritize PA, then weight management, and then medication adherence to mimic the emphasis in Phase II. Total weekly lesson time is 20-30 minutes. Patients retain access to lessons. They self-monitor calories, weight, moderate-to-vigorous physical activity, and medication adherence. Tracking data are seamlessly integrated into the system. They manually enter their medication adherence data and receive encouraging feedback on each of the behaviors the next week. Participants meeting responder criteria after 2 months will continue to receive the fully automated online program.
  Interventions: Behavioral: Fully Automated Online Program
- First Intervention: FAOP, Second Intervention: Low-Intensity Cardiac Rehabilitation (Experimental): Participants receive the fully automated online program for 2 months. Following their mid-intervention assessment, they are randomized to receive the low-intensity cardiac rehabilitation maintenance program. Patients are instructed to log in 3 times weekly to view lessons, sync their Fitbit data, and complete a home-based workout video. They track weight, PA, and medication adherence daily. Patients have access to an extensive CR resource library made and curated by the platform provider plus resources on maintaining heart healthy behaviors during Phase III created by the research team. They are reminded to log in if they log in less than twice weekly.
  Interventions: Behavioral: Fully Automated Online Program; Behavioral: Low-Intensity Cardiac Rehabilitation Maintenance Program
- First Intervention: FAOP, Second Intervention: High-Intensity Cardiac Rehabilitation (Experimental): Participants receive the fully automated online program intervention for 2 months. Following their mid-intervention assessment, they are randomized to receive the high-intensity cardiac rehabilitation maintenance program. Patients are instructed to log in 3 times weekly to view lessons, sync their Fitbit data, and complete a home-based workout video. They track weight, PA, and medication adherence daily and attend a once weekly virtual meeting with a CR case manager. Meetings are modeled after Phase II and focus on tailored exercise prescription, addressing cognitive, behavioral, and environmental adherence barriers, and support. Patients have access to an extensive CR resource library made and curated by the platform provider plus resources on maintaining heart healthy behaviors during Phase III created by the research team. They are reminded to log in (after they miss a login) if they log in less than twice weekly.
  Interventions: Behavioral: Fully Automated Online Program; Behavioral: High Intensity Cardiac Rehabilitation Maintenance Program

INTERVENTIONS:
Behavioral: Text Messaging — On 3 days/week they receive a text about 1 of the 3 behaviors (weight maintenance or loss, physical activity, and medication adherence) in randomized order with guidance for maintaining or improving these behaviors to reach program-provided goals. The system compares their last week's adherence to the responder criteria. They receive feedback praising adherence and instructions for a theory-driven behavioral strategy (e.g., stimulus control) to increase adherence. Feedback is tailored to the patient's adherence or existence of self-monitoring data.
  Arms: First Intervention: Text Messaging, Second Intervention: Continued Text Messaging; First Intervention: Text Messaging, Second Intervention: High-Intensity Cardiac Rehabilitation; First Intervention: Text Messaging, Second Intervention: Low-Intensity Cardiac Rehabilitation
Behavioral: Fully Automated Online Program — Patients receiving the fully automated online program will select a weight loss or a weight maintenance curriculum based on their goals. Patients will receive 8 weeks of fully automated lessons covering the 3 key behaviors: weight (management or loss), physical activity, and medication adherence. All 3 behaviors are discussed weekly, but the lessons first prioritize PA, then weight management, and then medication adherence to mimic the emphasis in Phase II. Total weekly lesson time is 20-30 minutes. Patients retain access to lessons. They self-monitor calories, weight, moderate-to-vigorous physical activity, and medication adherence. Tracking data are seamlessly integrated into the system. They manually enter their medication adherence data and receive encouraging feedback on each of the behaviors the next week.
  Arms: First Intervention: FAOP, Second Intervention: High-Intensity Cardiac Rehabilitation; First Intervention: FAOP, Second Intervention: Low-Intensity Cardiac Rehabilitation; First Intervention: Fully Automated Online Program (FAOP), Second Intervention: Continued FAOP
Behavioral: Low-Intensity Cardiac Rehabilitation Maintenance Program — Patients are instructed to log in 3 times weekly to view lessons, sync their Fitbit data, and complete a home-based workout video. They track weight, PA, and medication adherence daily. Patients have access to an extensive CR resource library made and curated by the platform provider plus resources on maintaining heart healthy behaviors during Phase III created by the research team. They are reminded to log in if they log in less than twice weekly.
  Arms: First Intervention: FAOP, Second Intervention: Low-Intensity Cardiac Rehabilitation; First Intervention: Text Messaging, Second Intervention: Low-Intensity Cardiac Rehabilitation
Behavioral: High Intensity Cardiac Rehabilitation Maintenance Program — Patients are instructed to log in 3 times weekly to view lessons, sync their Fitbit data, and complete a home-based workout video. They track weight, PA, and medication adherence daily and attend a once weekly virtual meeting with a CR case manager. Meetings are modeled after Phase II and focus on tailored exercise prescription, addressing cognitive, behavioral, and environmental adherence barriers, and support. Patients have access to an extensive CR resource library made and curated by the platform provider plus resources on maintaining heart healthy behaviors during Phase III created by the research team. They are reminded to log in if they log in less than twice weekly.
  Arms: First Intervention: FAOP, Second Intervention: High-Intensity Cardiac Rehabilitation; First Intervention: Text Messaging, Second Intervention: High-Intensity Cardiac Rehabilitation

SUMMARY:
The study is sponsored by the National Heart, Lung, and Blood Institute, which is part of the National Institutes of Health. We expect to enroll 400 subjects into this study. We will be recruiting research participants that are finishing or will finish cardiac rehabilitation soon. Participants belong to one or more groups of people who are less often studied in cardiac rehabilitation research, may have less access to a formal cardiac rehabilitation maintenance program, or they may especially benefit from additional support after cardiac rehabilitation ends. The main purposes of this study are to evaluate which treatments work the best after cardiac rehabilitation, which order to deliver the treatments in, and which treatments are as minimally burdensome as possible while still working well. This study will make two comparisons (one comparison between a set of low-intensity interventions and another between a set of higher-intensity interventions) to determine which produces the best behavioral adherence immediately after Phase II (outpatient) cardiac rehabilitation

DETAILED DESCRIPTION:
We will first test which of two automated online interventions ([A] a low-intensity text-messaging intervention of 3 weekly sets of text messages focused on encouragement and reminders about the key health behaviors for 2 months, or [B] a fully automated 2-month online program modeled on our previous research, consisting of interactive lessons, self-monitoring, and tailored feedback) serves as the best first-line intervention. The second test is which of two home-based cardiac rehabilitation (CR) maintenance interventions produces the best outcomes for non-responders to the initial interventions. Those who do not respond to the low-intensity interventions will be randomized to receive 3 months of either (C) low-intensity home-based CR, consisting of education and exercise prescription, or (D) high-intensity home-based online CR that includes education and exercise prescription plus case management. Adherence to the 3 targeted cardioprotective behaviors will be measured after Phase II completion (baseline), the initial low-touch interventions (at Month 3), after 3 more months of continued or new interventions (at Month 6), and 6-months of no-treatment follow-up (at Month 12). The primary outcome will be adherence to the 3 cardioprotective behaviors (physical activity, weight management, and medication adherence) measured together in the Sequential, Multiple Assignment, Randomized Trials (SMART) decision rule (responder status) and individually. Exploratory outcomes will be death, rehospitalization, and quality of life. The specific aims of this study are to: (1) Compare the 2 least intensive, online, intervention options (text message versus an automated online program) to determine which produces the best behavioral adherence immediately after Phase II CR; (2) Determine whether low- or high-intensity home-based CR (i.e., with or without case management) produces superior behavioral adherence after failure of initial low-intensity online intervention; (3) Finalize the adaptive treatment based on the results of the first two aims; and (4) [Exploratory Aim] Conduct a moderators analysis to test for differential effects within specific participant groups.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age or older
* Have completed at least 6 CR sessions
* Must enroll within 6 weeks of their final CR session
* BMI ≥27
* Own an internet-connected device
* Home internet access
* English proficiency
* Able to walk ≥1 block without stopping

Lastly, the participant MUST belong to ≥1 of the following groups or identities:

* Identifies as a woman
* Identifies as LGBTQIA+
* Identifies as a racial or ethnic minority
* Insecure transportation for medical appointments
* Self-reported trouble paying for healthcare needs (e.g., copays)
* Receive income-based subsidized benefits (e.g., state-funded health insurance for low-income residents)
* Reside in a small town or rural area per 2010 United States Department of Agriculture Rural-Urban Commuting Area zip code
* Low educational attainment (≤high school diploma)
* Low household income (less than twice the Federal Poverty Level) or meeting federal poverty guidelines per the National Committee on Vital and Health Statistics and the Department of Health and Human Services)

Exclusion Criteria:

* New York Heart Association Class IV heart failure
* Heart transplant in the last 5 months
* Left ventricular assist device in the last 4 months
* Physician diagnosis of dementia
* Physician prescription for 24 hours of oxygen therapy daily
* Coronary artery bypass surgery in the last 3 months
* Current dialysis
* Chronic gait or balance disturbances that would make unsupervised exercise unsafe
* Current pregnancy
* Report of conditions that the investigators believe would render them potentially unlikely to follow the protocol including terminal illness, active substance dependence, or other significant psychiatric problems that require inpatient hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-10-07 (Estimated); Study Completion 2030-03-29 (Estimated)

PRIMARY OUTCOMES:
Weight Management | From enrollment to the post-intervention assessment at 6 months
  Weight will be measured to the nearest 0.1 kg with a digital scale in light indoor clothing without shoes. Height will be measured to the nearest millimeter with standard stadiometer procedures; those without a recent (≤3 months) clinic height measurement will be sent a paper tape measure to be taped to a wall. BMI will be calculated (kg/m2). Local participants may come to the research center. Patients will be shipped a cellular-enabled scale to be used in the same location in their home for all assessments and will keep scales between assessments. Percent weight loss or management will be calculated as current weight/baseline weight.
Physical Activity | From enrollment to the post-intervention assessment at 6 months
  PA will be objectively measured over the 7-day assessment period via wearing the Fitbit on their wrist during waking hours. The Clinical Research Technologist can monitor device wear time during assessments and prompt participants to wear the device during their assessment period. Valid wear days will be defined as ≥600 min wear time during awake hours (e.g., 7am to 11pm; hours chosen with participant input) measured by non-zero heart rate measurements during that time and include patients with ≥4 valid days, including 1 weekend day. Fitbit allows researchers access to raw sensor data in 60 sec epochs via their API. Estimated mins/day spent in total PA and specific intensities of activities will be based on vertical axis counts/min thresholds primarily reflecting locomotor activity. The primary PA variable of interest will be MVPA mins/week.
Medication Adherence | From enrollment to the post-intervention assessment at 6 months
  Participants will complete a pill count of their total supply of common CVD medications. The medications will be counted at the assessment week beginning and end. Patients will complete the count twice; if the 2 do not agree, they will complete a third. The total number of pills will be recorded at each pill count. Percent adherence for each medication will be calculated as the difference between the baseline and end-of-treatment counts for that medication divided by the number of prescribed pills for that medication; this value will be multiplied by 100. Percent adherence per medication will be the difference between the baseline and end-of-treatment counts for that medication divided by the number of prescribed pills for that medication multiplied by 100. Percent adherence across medications will be the difference between baseline and end-of-treatment counts across all medications divided by the total number of prescribed pills for the 7-day period multiplied by 100.

SECONDARY OUTCOMES:
Hospitalizations | 12 months after enrollment
  Number of hospitalizations
Death | 12 months after enrollment
  Patients, the designated contacts, or the medical chart will provide information in the event that the participant has passed away since enrollment
Quality of life via the SF-36 | 12 months after enrollment
  Participants who are reached for the final assessment will complete a short survey form online or on the phone to measure their quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center of The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Due to the risk of re-identification in some communities, IPD will not be shared in this study.

REFERENCES:
- See also: Study Website — https://www.empowermestudy.com/